CLINICAL TRIAL: NCT03793751
Title: Effect of Intraoperative Dexmedetomidine Infusion on Early Postoperative Cognitive Dysfunction (POCD) in Geriatric Patients Undergoing Hip Surgery Under Spinal Anaesthesia
Brief Title: Effect of Intraoperative Dexmedetomidine on Early Postoperative Cognitive Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tata Main Hospital (Other)
Responsible Party: Principal Investigator, Dr.Deb Sanjay Nag, Consultant, Tata Main Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 201-26104-172-215441
Record Dates: First submitted 2018-12-30; First posted 2019-01-04 (Actual); Results first posted 2020-03-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a prospective, randomized, placebo-controlled, double-blind clinical trial. The patients will be recruited according to the inclusion criteria and will be distributed to one of the groups according to computer-generated random assignment. The personnel involved in the study, including statisticians, investigators, anaesthetists, surgeons and the patients will be blinded to the specific experimental scheme implementation Patients will be randomized into one of the two groups using a computer based random number generator. https://www.randomizer.org. All recordings would be performed by an anaesthesiologist blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEX Group (Experimental): Receiving Dexmedetomidine injection at a dose of 1 mcg/kg over 10 min, after Spinal Anaesthesia and before start of surgery, followed by a continuous infusion at a rate of 0.4 mcg/kg/h until the end of surgery.
  Interventions: Drug: Dexmedetomidine Injection
- CONTROL Group (Placebo Comparator): The Control Group will receive an equal volume placebo infusion of normal saline.
  Interventions: Drug: Dexmedetomidine Injection

INTERVENTIONS:
Drug: Dexmedetomidine Injection — Dexmedetomidine Injection at a dose of 1 mcg/kg over 10 min, after Spinal Anaesthesia and before start of surgery, followed by a continuous infusion at a rate of 0.4 mcg/kg/h until the end of surgery.
  Other Names: Normal Saline as placebo

SUMMARY:
This study will aim to identify the impact of Intraoperative dexmedetomidine infusion on POCD assessed by the Montreal Cognitive Assessment (MoCA) in geriatric patients above 60 years undergoing hip surgery under spinal anaesthesia.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is a common postoperative neurological complication in elderly. POCD is a subtle impairment of memory, concentration and information processing with clinical manifestations of delirium, anxiety, personality changes and impaired memory, which is associated with prolonged hospitalization, a reduced quality of life and an increase in morbidity and mortality. Dexmedetomidine is a highly selective α-2 adrenergic receptor agonist with a dose-dependent sedative hypnotic effect. It has also been reported that dexmedetomidine has a potential role in preventing POCD due to its neuroprotective effects both in vitro and in vivo.

Till date very few studies have analysed the impact of dexmedetomidine on early POCD. Even in the few available studies compared assessment of POCD using the Mini-Mental State Examination (MMSE) scores and found that MMSE have lower sensitivity for identifying Cognitive Dysfunction as compared to Montreal Cognitive Assessment (MoCA). The study would analyze the impact of Intraoperative Dexmedetomidine infusion on early Postoperative Cognitive Dysfunction (POCD) in geriatric patients above 60 years undergoing hip surgery under spinal anesthesia.

So this study will aim to identify the impact of Intraoperative dexmedetomidine infusion on POCD assessed by the Montreal Cognitive Assessment (MoCA) in geriatric patients above 60 years undergoing hip surgery under spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* American society of Anesthesiology (ASA) status of I-III
* Age between 60-75 years scheduled for elective hip surgery under spinal anesthesia

Exclusion Criteria:

* Patient not willing to be a part of the study
* Patients were aged <60 or >75 years
* Patients with accompanying medical conditions that may affect the level of consciousness, such as stroke, stupor or dementia, or patients with abnormalities in hepatic or renal function, electrolyte imbalance
* Patients suffering from preoperative bradycardia [heart rate (HR) <60 bpm] or hypotension [mean arterial blood pressure (MAP) <70 mmHg]
* Patients who had recently received a sedative or opioid drug
* Patients with a MoCA (Montreal Cognitive Assessment) score <26
* Patients with persistent hypotension and bradycardia intra-operatively even after giving Mephentermine will be excluded from the study

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Deb S Nag, MD, Principal Investigator — Tata Main Hospital
Locations (1):
- Dr.Deb Sanjay Nag, Jamshedpur, Jharkhand, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DEX Group: Dexmedetomidine injection at a dose of 1 mcg/kg over 10 min, after Spinal Anaesthesia and before start of surgery, followed by a continuous infusion at a rate of 0.4 mcg/kg/h until the end of surgery.
- CONTROL Group: The Control Group will receive placebo infusion of normal saline.
Period: Overall Study
Arm/Group | DEX Group | CONTROL Group
Started | 60 | 60
Completed | 60 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Geriatric patients of American Society of Anaesthesiology (ASA) status of I-III between 60-75 years scheduled for elective hip surgery under spinal anaesthesia.
Groups:
- Total: Total of all reporting groups
Arm/Group | DEX Group | CONTROL Group | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 41 | 40 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.28 (3.93) | 68.48 (4.96) | 68.38 (4.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 29 | 65
  Male | 24 | 31 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Indian | 60 | 60 | 120

OUTCOME MEASURES:

1. Primary Outcome: Number of Cases Developing POCD
Description: Number of cases developing POCD in the Dexmedetomidine Group as compared to the placebo group using the Montreal Cognitive Assessment (MoCA) test. The "Montreal Cognitive Assessment" (MoCA) test is a free assessment available at http://www.mocatest.org tool designed for quick screening for mild cognitive impairment. It is a one page, 30 point test done in approximately 10 min for assessment of attention, memory, abstraction, delayed recall and orientation, with total score of 30. MoCA range from zero to 30, with a score of 26 and higher generally considered normal. Scores below 26 were considered as Postoperative Cognitive Dysfunction.
Time Frame: 0-7 days
Measure: Count of Participants; unit: Participants
Arm/Group | DEX Group | CONTROL Group
Number analyzed (Participants) | 60 | 60
Participants | 10 | 21

2. Secondary Outcome: Systolic Blood Pressure
Description: Intraoperative Systolic Blood Pressure
Time Frame: Measured every 10 minutes upto 80 minutes, T0 as the initial reading.
Population: Intraoperative Systolic Blood Pressure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DEX Group | CONTROL Group
Number analyzed (Participants) | 60 | 60
mmHg
  T0 | 129.07 (13.5) | 125.4 (10.44)
  T1 | 130.78 (19.46) | 125.45 (10.81)
  T2 | 128.22 (13.78) | 127.48 (8.39)
  T3 | 126.22 (13.91) | 123.03 (8.6)
  T4 | 122.93 (13.47) | 119.1 (13.06)
  T5 | 117.71 (10.73) | 115.97 (11.43)
  T6 | 115.88 (10.65) | 113.5 (10.89)
  T7 | 117.71 (10.96) | 131.33 (15.31)
  T8 | 136.00 (5.29) | 155.00 (0)

3. Secondary Outcome: Diastolic Blood Pressure
Description: Intraoperative Diastolic Blood Pressure
Time Frame: Measured every 10 minutes upto 80 minutes, T0 as the initial reading.
Population: Diastolic Blood Pressure
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DEX Group | CONTROL Group
Number analyzed (Participants) | 60 | 60
mmHg
  T0 | 79.48 (9.38) | 80.40 (8.59)
  T1 | 78.92 (9.06) | 78.15 (11.19)
  T2 | 78.53 (7.61) | 80.17 (8.96)
  T3 | 75.15 (9.34) | 77.02 (10.28)
  T4 | 74.32 (8.44) | 72.77 (10.48)
  T5 | 72.69 (7.78) | 70.43 (11.96)
  T6 | 71.62 (7.35) | 68.38 (10.06)
  T7 | 71.79 (6.97) | 78 (7.81)
  T8 | 75.67 (5.51) | 90.00 (0)

4. Secondary Outcome: Heart Rate
Description: Intraoperative Heart Rate
Time Frame: Measured every 10 minutes upto 80 minutes, T0 as the initial reading.
Population: Intraoperative heart rate
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | DEX Group | CONTROL Group
Number analyzed (Participants) | 60 | 60
Beats/minute
  T0 | 75.00 (11.21) | 81.90 (7.09)
  T1 | 74.80 (11.37) | 82.02 (6.84)
  T2 | 79.8 (11.37) | 82.02 (6.81)
  T3 | 77.97 (11.27) | 82.65 (6.57)
  T4 | 76.32 (11.08) | 83.20 (6.18)
  T5 | 76.15 (10.57) | 84.00 (6.10)
  T6 | 74.76 (10.59) | 85.35 (6.15)
  T7 | 70.17 (10.46) | 86.67 (9.24)
  T8 | 69.33 (9.71) | 95.00 (0)

5. Secondary Outcome: Any Adverse Outcome
Description: Observation for any adverse effects
Time Frame: 0-7 days
Population: Insidence of adverse outcomes
Measure: Mean (Standard Deviation); unit: number of cases
Arm/Group | DEX Group | CONTROL Group
Number analyzed (Participants) | 60 | 60
number of cases | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: During the hospital admission upto 7 days after day of surgery
Description: Common adverse effects of dexmedetomidine: Hypotension, hypertension, bradycardia, dry mouth and nausea. Other reported adverse effects include fever, rigors, cyanosis, muscle weakness. It may lead to arrhythmias, AV Block, cardiac arrest, T-wave inversion, tachycardia, angina pectoris, pulmonary edema, bronchospasm, respiratory depression, syncope, neuropathy, paresthesia, paresis, hyperkalaemia, lactic acidosis and hyperglycaemia.
Arm/Group | DEX Group | CONTROL Group
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-01): https://cdn.clinicaltrials.gov/large-docs/51/NCT03793751/Prot_SAP_000.pdf